CLINICAL TRIAL: NCT01324869
Title: An Open-label, Randomized, Uncontrolled, Preliminary Clinical Study to Evaluate the Safety and Efficacy of KH902 Following Multiple Intravitreal Injection in Patients With Diabetic Macular Edema
Brief Title: Safety and Efficacy by Multiple Injection of KH902 in Patients With Diabetic Macular Edema (DME)
Acronym: Frontier-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Collaborators: University of Wisconsin, Madison (Other); Teaching and Research Office of Health Statistics, Fourth Military Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHSWKH902002
Record Dates: First submitted 2011-03-15; First posted 2011-03-29 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Diabetic Macular Edema
Keywords: KH902; Diabetic macular Edema; Intravitreal injection; Multiple injections; 20 patients; 0.5mg/eye/time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Patients will receive an intravitreal injection of 0.5mg KH902 in the study eye at the first month, following the fixed injection, patients will continue to receive injection of KH902 at the same dose on an as needed (PRN) dosing schedule based upon the monthly physician assessment of the need for re-treatment in accordance with pre-specified criteria.
  Interventions: Biological: KH902
- Group B (Experimental): Patients will receive continuously monthly intravitreal injections of 0.5 mg KH902 for 3 times in the study eye; following the initial 3-month fixed-dosing phase of the trial, patients will continue to receive injection of KH902 at the same dose on an as needed (PRN) dosing schedule based upon the monthly physician assessment of the need for re-treatment in accordance with pre-specified criteria.
  Interventions: Biological: KH902

INTERVENTIONS:
Biological: KH902 — Intravitreal injection of 0.5mg/eye/time KH902

SUMMARY:
This study is designed to access the safety and efficacy of multiple injections of KH902 in patients with Diabetic Macular Edema (DME).

DETAILED DESCRIPTION:
With improvement of our living standard, patients who suffered from Diabetes become more and more. As the investigators know, Diabetes can induce many ocular diseases leading to vision loss. And according to observations, DME is diagnosed as one main cause of vision loss in the patients with Diabetes.

As the results of many studies conducted previously, anti-VEGF drugs and anti-VEGF treatments show its effect and safety not only in treating AMD, but also in patients with DME. The new drug Recombinant Human VEGF Receptor-Fc Fusion Protein (KH902) is a gene fusion protein. The previous clinical trials of KH902 show that KH902 is effective and safe in inhibiting the growth, migration, pullulation of vascular endothelial cells and neovascularization induced by VEGF. Due to these positive results, the investigators prepare to conduct a clinical trial to assess the safety and efficacy with intravitreal injection of KH902 in patients with DME.

ELIGIBILITY:
Inclusion Criteria:

* Signed the Informed Consent Form and willing to comply with study procedures;
* 18 years old ≦ either gender ≦ 75 years old;
* Confirmed diagnosed with Type 1 diabetes or Type 2 diabetes based on the diabetes diagnosis criteria;
* Clinically significant DME:

  * Hard exudation within 500μm of the central foveal diameter accompanied with contiguous retina thickening;
  * The edema locates within 500μm of the central foveal diameter;
  * Retina thickening field > 1DD and within the 1DD central fovea.
* BCVA score of the study eyes between 78 and 19 letters, inclusively, and the BCVA score of fellow eyes ≥ 24 letters;
* Previous treatment of antidiabetic drugs within three months preceding the screening, and blood-glucose concentration is predicted to be unchanged and stable during the whole study.

Exclusion Criteria:

* Uncontrolled glaucoma in either eye;
* Currently active ocular inflammation or infection in either eye;
* Macular edema in the study eye was caused by other diseases rather than diabetes;
* Company with any other ocular conditions failing to prevent vision loss despite improving the macular edema;
* Any other ocular diseases which may cause macular edema or vision alteration during study phase;
* Retinal macular traction or macular epiretinal membrane in study eye;
* Refractive error equate or exceed 8 diopters of myopia in study eye
* Whole or regional retinal laser photocoagulation has been applied in study eye within 6 months preceding the screening;
* Previous anti-VEGF drug treatment in study eye;
* Intraocular or periocular injection of steroid drug within 6 months preceding the screening;
* Previous ophthalmologic operation within 3 months preceding the screening and/or planning to receive an ophthalmologic operation during the study.
* There is any potential for the study eye to receive the panretinal laser photocoagulation treatment during the study;
* Previous vitrectomy in study eye.
* Uncontrolled diabetes;
* Hypertensive patients with poorly controlled blood pressure;
* Uncontrolled systemic infectious diseases;
* Systemic immune diseases;
* History of allergy;
* Any uncontrolled clinical disorders;
* Pregnant or nursing women;
* Adopt one or more adequate contraception methods.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence rate of adverse event | up to 12 months
  To evaluate the safety of multiple intravitreal injection of KH902 to treat DME.

SECONDARY OUTCOMES:
Change from Baseline in BCVA | at the end of month 3 and the end of month 12
  To evaluate the efficacy of multiple intravitreal injection of KH902 of each group.

CONTACTS AND LOCATIONS:
Overall Officials: Xun Xu, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Lun De Luo, Study Director — Chengdu Kanghong Biotech Co., Ltd.
Locations (1):
- Shanghai First People's Hospital, Shanghai, China